CLINICAL TRIAL: NCT06887946
Title: Effectiveness of Medical Coaching in Enhancing Periodontal Health and Lifestyle: A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Medical Coaching in Enhancing Periodontal Health and Lifestyle
Acronym: MCOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Medical Coaching in Perio
Record Dates: First submitted 2025-03-19; First posted 2025-03-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Periodontitis
Keywords: Medical Coaching; Periodontitis; Stress; gingival health
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Couching (Experimental): MCOH group (n=32) . The baseline assessments included periodontal status, PCR, GBI (describe the achronym) and a systematic questionnaire on lifestyle factors (smoking, alcohol, food, exercise, sleep, and stress). The intervention group received tailored MCOH sessions that comprised goal-setting, emotional hurdle assessment and action planning, whereas the control group received conventional OHI.
  Interventions: Other: Medical couching and traditional
- control group (Other): Control group (n=32.)Control group received traditional OHI using the tell-show-do method, which was personalized based on the individual PCR and GBI. The recommendations were tailored to each participant, based on personalized instructions to improve plaque control, decrease of gingival inflammation and facilitate optimal patient compliance, contributing to oral hygiene performance.
  Interventions: Other: Medical couching and traditional

INTERVENTIONS:
Other: Medical couching and traditional — The control group received traditional OHI using the tell-show-do method, which was personalized based on the individual PCR and GBI. The recommendations were tailored to each participant, based on personalized instructions to improve plaque control, decrease of gingival inflammation and facilitate optimal patient compliance, contributing to oral hygiene performance.
  The intervention group was actively engaged in an iterative, collaborative process, based on the following steps:
  Definition of the goals of oral hygiene and lifestyle styles according to the SMART model (Specific, Measurable, Achievable, Realistic, Timely):

SUMMARY:
Periodontitis is a chronic inflammatory disease that adversely influences the supporting tissues of the teeth. It is primarily characterized by the accumulation of bacterial plaque and the host immune response. Traditional periodontal therapy emphasizes the central roles of both oral hygiene education and risk factor management; however, maintaining a long-term optimal behavioral compliance remains challenging.

The purpose of this Randomized Controlled Trial is to assess how effective is Medical Coaching on Oral Health (MCOH) in improving plaque control (PCR) and gingival health (GBI) in patients with periodontitis after one month, in comparison to traditional oral hygiene instructions (OHI).

DETAILED DESCRIPTION:
The baseline assessments included periodontal status, PCR, GBI (describe the achronym) and a systematic questionnaire on lifestyle factors (smoking, alcohol, food, exercise, sleep, and stress). The intervention group received tailored MCOH sessions that comprised goal-setting, emotional hurdle assessment and action planning, whereas the control group received conventional OHI.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis Patients

Exclusion Criteria:

* Patients who do not wish to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Plaque Control Record (PCR) . | 30 days
  The percentage value was calculated as follows: Number of surfaces with plaque / Total number of surfaces examined × 100. The lower the percentage, the better the plaque control; the higher the percentage, the worse the oral hygiene.
Gingival Bleeding Index (GBI) | 30 days
  The calculation to the GBI was as follows: number of bleeding sites/number of evaluated sites ×100. obtain the percentage value was as follows: number of bleeding sites/number of evaluated sites ×100

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis Dr, DDS, Principal Investigator — University of Bari Aldo Moro
Locations (1):
- Anna Antonacci, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antonacci A, D'Albis G, Bartolomeo N, Agneta MT, Abbinante A, Marini L, Pilloni A, Capodiferro S. Effectiveness of Medical Coaching in Enhancing Periodontal Health and Lifestyle: A Clinical Trial. Oral Dis. 2026 Jan 7. doi: 10.1111/odi.70183. Online ahead of print. PMID 41501894